CLINICAL TRIAL: NCT02568488
Title: The Effect of Metformin on Serum Insulin, Androgens and AMH in PCOS Patients
Brief Title: The Effect of Metformin on Different Hormones in PCOS Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ahmed Maged (Other)
Responsible Party: Sponsor-Investigator, Ahmed Maged, Assistant professor, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 138
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- metformin (Experimental): PCOS women receiving metformin 850 mg orally twice daily over a period of 6 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg orally twice daily for 6 months
  Other Names: glucophage

SUMMARY:
Forty eight PCOS patients were included . The diagnosis of PCOS was made based on the three criteria set by the Rotterdam Consensus meeting definition of PCOS (ESHRE, ASRM, 2004). The criteria were as follows:

1. history of chronic anovulation defined as cycle length > 35 days, or less than 9 cycles per year or amenorrhoea (cycle length > 12wks),
2. infertility with hirsutism or acne or elevation of one or more of serum androgen levels
3. ultrasonographic findings of polycystic ovaries ( increased ovarian volume, more than eight follicles in an ovary ranging from 2-10mm).

the studied subjects were to receive metformin 850 mg twice daily over a period of 6 months. Blood samples were collected at the start of the study, before receiving metformin, where baseline serum insulin (fasting and 2 hr postprandial), sex hormone binding globulin (SHBG) , total and free testosterone, Dihydroepiandrostenedione sulphate (DHEAS) and Antimullerian Hormone (AMH) were obtained before starting metformin. Blood samples were collected at 3 and 6 months respectively of metformin treatment , to asses its effect on serum levels of the previously mentioned hormonal parameters.

DETAILED DESCRIPTION:
Forty eight PCOS patients attending the OBGYN clinic at kasr al aini were included in the study. The diagnosis of PCOS was made based on the three criteria set by the Rotterdam Consensus meeting definition of PCOS (ESHRE, ASRM, 2004). The criteria were as follows:

1. history of chronic anovulation defined as cycle length > 35 days, or less than 9 cycles per year or amenorrhoea (cycle length > 12wks),
2. infertility with hirsutism or acne or elevation of one or more of serum androgen levels
3. ultrasonographic findings of polycystic ovaries ( increased ovarian volume, more than eight follicles in an ovary ranging from 2-10mm).

the studied subjects were to receive metformin 850 mg twice daily over a period of 6 months. Blood samples were collected at the start of the study, before receiving metformin, where baseline serum insulin (fasting and 2 hr postprandial), sex hormone binding globulin (SHBG) , total and free testosterone, Dihydroepiandrostenedione sulphate (DHEAS) and Antimullerian Hormone (AMH) were obtained before starting metformin. Blood samples were collected at 3 and 6 months respectively of metformin treatment , to asses its effect on serum levels of the previously mentioned hormonal parameters.

The effect of metformin on PCOS patients regarding its clinical and radiological parameters was also assessed. Each patient was asked to keep a diary of her menstrual periods over the study period; to elicit if there could be an effect by metformin on the regulation of menstrual cycles secondary to improvement of ovarian function as a result of improving insulin resistance in such patients. The effect of metformin on ovarian morphology by ultrasound was also assessed at baseline, 3months and 6 months of the study period; ovarian volume and number of follicles was noted down at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Non pregnant PCOS patients .
* The diagnosis of PCOS was made based on the three criteria set by the Rotterdam Consensus meeting definition of PCOS (ESHRE, ASRM, 2004). The criteria were as follows:

  1. history of chronic anovulation defined as cycle length > 35 days, or less than 9 cycles per year or amenorrhoea (cycle length > 12wks),
  2. infertility with hirsutism or acne or elevation of one or more of serum androgen levels
  3. ultrasonographic findings of polycystic ovaries ( increased ovarian volume, more than eight follicles in an ovary ranging from 2-10mm).

Exclusion Criteria:

* those with prior history of glucose intolerance,
* history of gestational diabetes,
* NIDDM patients,
* cushing's syndrome,
* thyroid dysfunction,
* hyperprolactinemia,
* congenital adrenal hyperplasia
* patients on prolonged corticosteroid course, or other medications that alter the hormonal or metabolic profile; including PCOS patients who were on OCPs or cyclic progestagens

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
hormonal changes | Change from Baseline at 3 and 6 months
  total and free testosterone

SECONDARY OUTCOMES:
serum insulin levels | Change from Baseline at 3 and 6 months
  serum insulin (fasting and 2 hr postprandial)
ovarian morphology | Change from Baseline at 3 and 6 months
  ovarian volume and number of follicles
sex hormone binding globulin (SHBG) | Change from Baseline at 3 and 6 months
Antimullerian Hormone (AMH) | Change from Baseline at 3 and 6 months
Dihydroepiandrostenedione sulphate (DHEAS) | Change from Baseline at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school